CLINICAL TRIAL: NCT07364110
Title: Comparison of High Intensity Laser Therapy (HILT) and Extracorporeal Shock Wave Therapy (ESWT) for the Treatment of Plantar Flexor Spasticity in Post-Stroke Patients
Brief Title: The Effectiveness of Laser and Extracorporeal Shock Wave Therapy in Resolving Ankle Muscle Spasm in Stroke Patients.
Acronym: spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, SAMİ KÜÇÜKŞEN, Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/454; 221518007 (Other Grant/Funding Number: Necmettin Erbakan University, Scientific Research Projects)
Record Dates: First submitted 2025-12-28; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2021-05

CONDITIONS: Stroke Gait Rehabilitation
Keywords: stroke; spasticity; equinus deformity; extracorporeal shock wave therapy; high-intensity laser therapy
MeSH Terms: conditions — Stroke; Muscle Spasticity; Equinus Deformity | interventions — Exercise; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rehabilitation-only group (Placebo Comparator): All participants received a standardized rehabilitation program consisting of 1-hour sessions, 5 days per week, for 3 consecutive weeks. The program included:
  * Range of motion and stretching exercises targeting the hamstrings, rectus femoris, and ankle plantar flexors;
  * Strengthening exercises for hip flexors, hip extensors, knee extensors, hamstrings, ankle plantar flexors, and trunk muscles;
  * Gait training, postural exercises, balance training, transfer training, and endurance exercises, all performed under the supervision of a physiotherapist.
  Interventions: Procedure: Rehabilitation Protocol
- ESWT plus rehabilitation group (Experimental): Participants in the ESWT group received ESWT once weekly for 3 consecutive weeks (total of 3 sessions), in addition to the rehabilitation program. ESWT was applied to the gastrocnemius muscle belly in the prone position using a Starz Medical Masterpuls MP100 device, with the following parameters: frequency 5 Hz, energy flux density 0.340 mJ/mm², 2000 pulses, and a 15-mm applicator.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- HILT plus rehabilitation group (Experimental): In addition to the rehabilitation program, participants in the HILT group received HILT three times per week for 3 consecutive weeks (total of 9 sessions). Each session lasted 4 minutes. HILT was applied to the gastrocnemius muscle belly in the prone position using longitudinal movements, with an energy density of 50 J/cm² and output power of 5 W in biostimulatory mode, using a BTL-6000 High-Intensity Laser device.
  Interventions: Device: High-Intensity Laser Therapy (HILT)

INTERVENTIONS:
Procedure: Rehabilitation Protocol — All participants received a standardized rehabilitation program consisting of 1-hour sessions, 5 days per week, for 3 consecutive weeks. The program included:
  * Range of motion and stretching exercises targeting the hamstrings, rectus femoris, and ankle plantar flexors;
  * Strengthening exercises for hip flexors, hip extensors, knee extensors, hamstrings, ankle plantar flexors, and trunk muscles;
  * Gait training, postural exercises, balance training, transfer training, and endurance exercises, all performed under the supervision of a physiotherapist
  Other Names: Exercise
  Arms: Rehabilitation-only group
Device: Extracorporeal Shock Wave Therapy (ESWT) — Participants in the ESWT group received ESWT once weekly for 3 consecutive weeks (total of 3 sessions), in addition to the rehabilitation program. ESWT was applied to the gastrocnemius muscle belly in the prone position using a Starz Medical Masterpuls MP100 device, with the following parameters: frequency 5 Hz, energy flux density 0.340 mJ/mm², 2000 pulses, and a 15-mm applicator.
  Other Names: 2
  Arms: ESWT plus rehabilitation group
Device: High-Intensity Laser Therapy (HILT) — In addition to the rehabilitation program, participants in the HILT group received HILT three times per week for 3 consecutive weeks (total of 9 sessions). Each session lasted 4 minutes. HILT was applied to the gastrocnemius muscle belly in the prone position using longitudinal movements, with an energy density of 50 J/cm² and output power of 5 W in biostimulatory mode, using a BTL-6000 High-Intensity Laser device.
  Other Names: 3
  Arms: HILT plus rehabilitation group

SUMMARY:
Stroke is one of the leading causes of long-term disability worldwide. Spasticity (muscle spasm) is a common and disabling consequence of stroke. Lower extremity spasticity significantly compromises postural control, balance, and gait performance. Patients with spasticity demonstrate greater difficulty in standing and walking compared with non-spastic stroke survivors.

Management of spasticity includes physical therapy modalities, exercise programs, orthoses, and pharmacological agents. In recent years, novel noninvasive treatment modalities including extracorporeal shock wave therapy (ESWT), and low- and high-intensity laser therapy (HILT) have been investigated for spasticity management however, robust evidence remains limited.

ESWT is a treatment method applied by focusing high-pressure sound waves produced outside the body on the desired area of the body using a steel-tipped applicator. Patients can resume their daily activities immediately after a treatment session lasting between 5-20 minutes. Scientific researches have demonstrated that ESWT is a safe and effective modality for reducing upper and lower extremity spasticity after stroke.

HILT is a a non-invasive, advanced therapeutic approach that utilizes high-intensity laser technology to promote healing and alleviate pain. It has been widely used in musculoskeletal disorders and generally well tolerated without significant adverse effects. Previous studies suggest that laser application to spastic muscles after stroke may reduce spasticity and pain.

The present study aimed to investigate and compare the effects of ESWT and HILT applied to the calf muscles on spasticity and functional gait parameters only with clinical examination methods in patients with stroke.

DETAILED DESCRIPTION:
Stroke is defined as an acute episode of focal dysfunction of the brain, retina, or spinal cord lasting longer than 24 hours, or of any duration if imaging or autopsy demonstrates focal infarction or hemorrhage relevant to the symptoms.

Stroke is one of the leading causes of mortality, long-term disability, and socioeconomic burden worldwide. Although approximately 88% of patients survive a stroke, a substantial proportion experience persistent impairments that limit independent living and participation in daily activities.

Spasticity is a common and disabling consequence of stroke and is defined as a motor disorder characterized by a velocity-dependent increase in tonic stretch reflexes resulting from abnormal intra-spinal processing of primary afferent input. It arises from impaired reflex modulation and leads to secondary changes in muscle tissue such as increased stiffness, fibrosis, and muscle atrophy. Post-stroke spasticity affects approximately 30% of patients and may develop at variable time points following stroke onset.

Lower extremity spasticity significantly compromises postural control, balance, and gait performance. Patients with spasticity demonstrate greater difficulty in standing and walking compared with non-spastic stroke survivors. Among lower limb muscles, the gastrocnemius medialis is most frequently affected, and its involvement is strongly associated with impaired gait mechanics and reduced walking efficiency.

Management of spasticity includes physical therapy modalities, comprehensive neurorehabilitation programs, orthoses, pharmacological agents, and surgical interventions. Stretching exercises constitute the cornerstone of rehabilitation, aiming to improve the viscoelastic properties of the muscle-tendon unit and prevent fixed contractures.

Systemic pharmacological treatment is generally reserved for generalized spasticity, whereas focal spasticity is preferably managed with local treatments such as phenol, alcohol, or botulinum toxin type A injections.

In recent years, novel noninvasive treatment modalities including extracorporeal shock wave therapy, low- and high-intensity laser therapy, dry needling, and therapeutic ultrasound have been investigated for spasticity management; however, robust evidence remains limited.

Laser therapy is a noninvasive modality that induces biological effects at the cellular and tissue levels depending on wavelength, energy density, and power. Both low-intensity and high-intensity laser therapies have been widely used in musculoskeletal disorders and are generally well tolerated with a low incidence of adverse effects. Previous studies suggest that laser application to spastic muscles after stroke may reduce spasticity and pain while improving joint range of motion and muscle endurance.

Extracorporeal shock wave therapy consists of short-duration, high-pressure acoustic pulses transmitted to biological tissues. Radial ESWT delivers lower energy and peak pressure compared with focused ESWT, with therapeutic penetration up to approximately 3.5 cm. Proposed mechanisms of action include nitric oxide release, neuromodulation, axonal regeneration, enhancement of vascular endothelial growth factor activity, and increased expression of neurotrophins, leading to improved neural and muscular function.

Systematic reviews and meta-analyses have demonstrated that ESWT is a safe and effective modality for reducing upper and lower extremity spasticity after stroke, with significant reductions in MAS scores reported immediately after treatment and at short-term follow-up.

Despite improvements in muscle tone, the impact of spasticity treatments on functional gait outcomes remains insufficiently established. Therefore, the development of novel treatment strategies is necessary to optimize functional recovery in stroke survivors.

The present study aimed to investigate and compare the effects of ESWT and HILT applied to the gastrocnemius muscle on plantar flexor spasticity and functional gait parameters in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever stroke;
2. At least 3 months elapsed since stroke onset;
3. Age ≥18 years;
4. Presence of ankle plantar flexor spasticity graded 1-3 on the Modified Ashworth Scale (MAS);
5. Ability to ambulate independently or under supervision with or without assistive devices/orthoses;
6. Sufficient cognitive capacity to understand and follow test instructions

Exclusion Criteria:

* Fixed ankle contracture (peak ankle dorsiflexion <0° with the knee in extension);
* Current use of antispastic medications or a history of botulinum toxin injection within the previous 4 months;
* Any orthopedic, rheumatologic, neurologic, cardiovascular, or visual comorbidity other than stroke that could affect gait;
* Insufficient cognitive function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  Plantar flexor spasticity was assessed using the Modified Ashworth Scale (MAS), a widely used clinical instrument for evaluating resistance to passive movement. The MAS is employed to quantify increases in muscle tone and grades spasticity on an ordinal scale ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates rigidity of the affected limb in flexion or extension.

SECONDARY OUTCOMES:
Ankle Range of Motion (ROM) | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  Ankle dorsiflexion range of motion was measured using a standard goniometer, with the hip and knee positioned at 90° of flexion. The normal range of ankle dorsiflexion is considered to be approximately 20 degrees.
Fugl-Meyer Lower Extremity Assessment (FM-LE) | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  The Fugl-Meyer Lower Extremity Assessment (FM-LE) is a standardized and validated tool used to quantify motor recovery following stroke. It evaluates motor impairments of the lower extremity as well as postural control. The FM-LE consists of 14 items assessing movements of the hip, knee, and ankle. Each item is scored on a 3-point ordinal scale ranging from 0 (no active movement) to 2 (normal movement), with a maximum possible score of 28 points (range: 0-28). Higher scores indicate better motor function and greater recovery.
Timed Up and Go Test (TUG) | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  The Timed Up and Go Test (TUG) is a functional mobility assessment used to evaluate balance, walking ability, and fall risk in older adults and individuals with neurological disorders. The test measures the time required for an individual to stand up from a chair, walk three meters, turn around, walk back, and sit down. Longer completion times indicate poorer functional performance. A TUG time of 20 seconds or more is associated with reduced physical performance and an increased risk of falls.
10-Meter Walk Test | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  The 10-Meter Walk Test is a performance-based measure used to assess gait speed, expressed in meters per second, over a short distance. It is commonly utilized to evaluate functional mobility, gait efficiency, and balance. In individuals with stroke, walking speeds below 0.7 m/s are associated with an increased risk of falls, hospitalization, and dependency in daily activities.
Berg Balance Scale (BBS) | Baseline, at 3 weeks (end of intervention), and at 12 weeks (follow-up).
  The Berg Balance Scale (BBS) is a clinical assessment tool used to objectively evaluate static and dynamic balance through a series of functional tasks, including sitting to standing, standing under varying sensory and base-of-support conditions, reaching, turning, and stepping. The scale consists of 14 items, each scored on a 5-point scale from 0 to 4, yielding a maximum total score of 56 points. Higher scores indicate better balance performance, whereas lower scores are associated with an increased risk of falls. A score of 49 or below is considered indicative of fall risk in individuals with stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Meram Medical School, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication- ending 2 years after the publication of results
Access Criteria: Journal editors or reviewers may request this information from the corresponding author's email address if they deem it necessary.

REFERENCES:
- [Result] Mizuta N, Hasui N, Nakatani T, Takamura Y, Fujii S, Tsutsumi M, Taguchi J, Morioka S. Walking characteristics including mild motor paralysis and slow walking speed in post-stroke patients. Sci Rep. 2020 Jul 16;10(1):11819. doi: 10.1038/s41598-020-68905-3. PMID 32678273
- [Result] Bushnell C, Bettger JP, Cockroft KM, Cramer SC, Edelen MO, Hanley D, Katzan IL, Mattke S, Nilsen DM, Piquado T, Skidmore ER, Wing K, Yenokyan G. Chronic Stroke Outcome Measures for Motor Function Intervention Trials: Expert Panel Recommendations. Circ Cardiovasc Qual Outcomes. 2015 Oct;8(6 Suppl 3):S163-9. doi: 10.1161/CIRCOUTCOMES.115.002098. PMID 26515205
- [Result] Wade DT. Measurement in neurological rehabilitation. Curr Opin Neurol Neurosurg. 1992 Oct;5(5):682-6. PMID 1392142
- [Result] Blum L, Korner-Bitensky N. Usefulness of the Berg Balance Scale in stroke rehabilitation: a systematic review. Phys Ther. 2008 May;88(5):559-66. doi: 10.2522/ptj.20070205. Epub 2008 Feb 21. PMID 18292215
- [Result] Bohannon RW. Reference values for the timed up and go test: a descriptive meta-analysis. J Geriatr Phys Ther. 2006;29(2):64-8. doi: 10.1519/00139143-200608000-00004. PMID 16914068
- [Result] Amelio E, Manganotti P. Effect of shock wave stimulation on hypertonic plantar flexor muscles in patients with cerebral palsy: a placebo-controlled study. J Rehabil Med. 2010 Apr;42(4):339-43. doi: 10.2340/16501977-0522. PMID 20358168
- [Result] Troncati F, Paci M, Myftari T, Lombardi B. Extracorporeal Shock Wave Therapy reduces upper limb spasticity and improves motricity in patients with chronic hemiplegia: a case series. NeuroRehabilitation. 2013;33(3):399-405. doi: 10.3233/NRE-130970. PMID 23949081
- [Result] Starosta M, Marek K, Redlicka J, Miller E. Extracorporeal Shockwave Treatment as Additional Therapy in Patients with Post-Stroke Spasticity of Upper Limb-A Narrative Review. J Clin Med. 2024 Mar 30;13(7):2017. doi: 10.3390/jcm13072017. PMID 38610782
- [Result] Moon SW, Kim JH, Jung MJ, Son S, Lee JH, Shin H, Lee ES, Yoon CH, Oh MK. The effect of extracorporeal shock wave therapy on lower limb spasticity in subacute stroke patients. Ann Rehabil Med. 2013 Aug;37(4):461-70. doi: 10.5535/arm.2013.37.4.461. Epub 2013 Aug 26. PMID 24020026
- [Result] Li TY, Chang CY, Chou YC, Chen LC, Chu HY, Chiang SL, Chang ST, Wu YT. Effect of Radial Shock Wave Therapy on Spasticity of the Upper Limb in Patients With Chronic Stroke: A Prospective, Randomized, Single Blind, Controlled Trial. Medicine (Baltimore). 2016 May;95(18):e3544. doi: 10.1097/MD.0000000000003544. PMID 27149465
- [Result] Daliri SS, Forogh B, Emami Razavi SZ, Ahadi T, Madjlesi F, Ansari NN. A single blind, clinical trial to investigate the effects of a single session extracorporeal shock wave therapy on wrist flexor spasticity after stroke. NeuroRehabilitation. 2015;36(1):67-72. doi: 10.3233/NRE-141193. PMID 25547767
- [Result] Guo P, Gao F, Zhao T, Sun W, Wang B, Li Z. Positive Effects of Extracorporeal Shock Wave Therapy on Spasticity in Poststroke Patients: A Meta-Analysis. J Stroke Cerebrovasc Dis. 2017 Nov;26(11):2470-2476. doi: 10.1016/j.jstrokecerebrovasdis.2017.08.019. Epub 2017 Sep 13. PMID 28918085
- [Result] Dymarek R, Ptaszkowski K, Slupska L, Halski T, Taradaj J, Rosinczuk J. Effects of extracorporeal shock wave on upper and lower limb spasticity in post-stroke patients: A narrative review. Top Stroke Rehabil. 2016 Aug;23(4):293-303. doi: 10.1080/10749357.2016.1141492. Epub 2016 Feb 17. PMID 27077981
- [Result] Radinmehr H, Nakhostin Ansari N, Naghdi S, Olyaei G, Tabatabaei A. Effects of one session radial extracorporeal shockwave therapy on post-stroke plantarflexor spasticity: a single-blind clinical trial. Disabil Rehabil. 2017 Mar;39(5):483-490. doi: 10.3109/09638288.2016.1148785. Epub 2016 Mar 13. PMID 26971745
- [Result] das Neves MF, Dos Reis MC, de Andrade EA, Lima FP, Nicolau RA, Arisawa EA, Andrade AO, Lima MO. Effects of low-level laser therapy (LLLT 808 nm) on lower limb spastic muscle activity in chronic stroke patients. Lasers Med Sci. 2016 Sep;31(7):1293-300. doi: 10.1007/s10103-016-1968-x. Epub 2016 May 31. PMID 27299571
- [Result] Song HJ, Seo HJ, Lee Y, Kim SK. Effectiveness of high-intensity laser therapy in the treatment of musculoskeletal disorders: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Dec;97(51):e13126. doi: 10.1097/MD.0000000000013126. PMID 30572425
- [Result] Chen B, Yang T, Liao Z, Sun F, Mei Z, Zhang W. Pathophysiology and Management Strategies for Post-Stroke Spasticity: An Update Review. Int J Mol Sci. 2025 Jan 5;26(1):406. doi: 10.3390/ijms26010406. PMID 39796261
- [Result] Kesar TM, Perumal R, Reisman DS, Jancosko A, Rudolph KS, Higginson JS, Binder-Macleod SA. Functional electrical stimulation of ankle plantarflexor and dorsiflexor muscles: effects on poststroke gait. Stroke. 2009 Dec;40(12):3821-7. doi: 10.1161/STROKEAHA.109.560375. Epub 2009 Oct 15. PMID 19834018
- [Result] Thibaut A, Chatelle C, Ziegler E, Bruno MA, Laureys S, Gosseries O. Spasticity after stroke: physiology, assessment and treatment. Brain Inj. 2013;27(10):1093-105. doi: 10.3109/02699052.2013.804202. Epub 2013 Jul 25. PMID 23885710
- [Result] Young RR. Spasticity: a review. Neurology. 1994 Nov;44(11 Suppl 9):S12-20. PMID 7970006
- [Result] Jan S, Arsh A, Darain H, Gul S. A randomized control trial comparing the effects of motor relearning programme and mirror therapy for improving upper limb motor functions in stroke patients. J Pak Med Assoc. 2019 Sep;69(9):1242-1245. PMID 31511706
- [Result] Hankey GJ. Stroke. Lancet. 2017 Feb 11;389(10069):641-654. doi: 10.1016/S0140-6736(16)30962-X. Epub 2016 Sep 13. PMID 27637676
- [Result] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265